CLINICAL TRIAL: NCT04623892
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerance and Pharmacokinetics of TQB2618 Injection in Subjects With Advanced Solid Tumors
Brief Title: A Study to Evaluate the Tolerance and Pharmacokinetics of TQB2618 Injection in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-I-01
Record Dates: First submitted 2020-11-08; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-02

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2618 (Experimental): TQB2618 administered intravenously (IV) on Day 1 of each 21-day.
  Interventions: Drug: TQB2618 injection

INTERVENTIONS:
Drug: TQB2618 injection — TQB2618 administered intravenously (IV) on Day 1 of each 21-day. The established dose of TQB2618 is diluted to 100 m with normal saline [0.9% (w/v) sodium chloride solution], and the infusion time is 60 ± 10 min.

SUMMARY:
TQB2618 is a TIM-3 receptor monoclonal antibody that binds to the extracellular domain of TIM-3 outside the cell to block the binding of TIM-3 to its ligand, thereby inhibiting the downstream signal transduction of TIM-3 and deactivating TIM-3 Inhibition of immune cells. The purpose of this study was to evaluate the safety, tolerability, pharmacokinetic parameters and antitumor effects of TQB2618 injection in subjects with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed as advanced malignant solid tumors and have failed standard treatments or lack effective treatments; 2. 18-75 years old; Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1; Life expectancy ≥12 weeks; 3. Has at least one measurable lesion; 4. The function of main organs is normal; 5. Female patients of childbearing age must be negative in serum or urine HCG within 7 days before enrollment in the study, and must be non-lactating; patients should agree to use contraceptive measures during the study period and within 6 months after the end of the study period; 6. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has Autoimmune disease; 2. Has received allogeneic bone marrow transplantation or solid organ transplantation; 3. Has brain disease or brain metastases; 4. Has cavity effusion; 5. Has cardiovascular diseases; 6. Has immunodeficiency diseases; 7. Has liver disease; 8. Has infection; 9. Has diabetes; 10. Has a history of psychotropic drug abuse or have a mental disorder; 11. Have a history of severe allergy to macromolecular drugs or allergy to known components of TQB2618 injection; 12. Has other malignant tumors within 2 years before the first medication; 13. Has received other anti-cancer drugs or anti-cancer treatments, or major surgical operations within 4 weeks before the first medication; 14. Has received any live vaccines or vaccines to prevent infectious diseases within 4 weeks before the first medication; 15. Has received local radiotherapy within 1 week before the first medication; 16. Toxicity (excluding hair loss) caused by previous anti-tumor therapy that has not recovered to CTC AE V5.0 level 1 or below; 17. Has major wound, severe ulcer or fracture that has not healed before 1 day before the first medication; 18. Has used systemic hormones, immune agonists, inhibitors, and regulators before 1 day before the first medication; 19. According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Baseline up to 28 days
  MTD was defined as the dose in which more than 2 of up to 6 patients developed a DLT.

SECONDARY OUTCOMES:
Tmax | Pre-dose, 30 minutes, 4 hours, 8 hours, 24 hours, 48 hours, 144 hours, 312 hours post-dose on day 1 and day 43; Pre-dose, 30 minutes post-dose within the second, fourth, sixth and eighth cycles. Each cycle is 21 days.
  To characterize the pharmacokinetics of TQB2618 by assessment of time to reach maximum plasma concentration.
Cmax | Pre-dose, 30 minutes, 4 hours, 8 hours, 24 hours, 48 hours, 144 hours, 312 hours post-dose on day 1 and day 43; Pre-dose, 30 minutes post-dose within the second, fourth, sixth and eighth cycles. Each cycle is 21 days.
  Cmax is the maximum plasma concentration of TQB2618 or metabolite(s).
t1/2 | Pre-dose, 30 minutes, 4 hours, 8 hours, 24 hours, 48 hours, 144 hours, 312 hours post-dose on day 1 and day 43; Pre-dose, 30 minutes post-dose within the second, fourth, sixth and eighth cycles. Each cycle is 21 days.
  t1/2 is time it takes for the blood concentration of TQB2618 injection or metabolite(s) to drop by half.
AUC0-t | Pre-dose, 30 minutes, 4 hours, 8 hours, 24 hours, 48 hours, 144 hours, 312 hours post-dose on day 1 and day 43; Pre-dose, 30 minutes post-dose within the second, fourth, sixth and eighth cycles. Each cycle is 21 days.
  To characterize the pharmacokinetics of TQB2618 by assessment of area under the plasma concentration time curve from zero to infinity.
Receptor occupation (RO) | Pre-dose, 30 minutes, 4 hours, 8 hours, 24 hours, 48 hours, 144 hours, 312 hours post-dose on day 1 and day 43; Pre-dose, 30 minutes post-dose within the second, fourth, sixth and eighth cycles. Each cycle is 21 days.
  Receptor occupation of TIM-3 after single and multiple doses
Overall response rate (ORR) | Up to 48 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Progression-free survival (PFS) | Up to 48 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Disease control rate（DCR） | Up to 48 weeks
  Percentage of participants achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Duration of response (DOR) | Up to 48 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of The University of Chinese Academy of Sciences, Hangzhou, Zhejiang, China